CLINICAL TRIAL: NCT01794884
Title: Intravenous Supplementation of Glutamine Preoperatively for Cardiac Function and Recovery Improvement in Adult Accepting Cardiosurgery: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Validity Study of Glutamine to Improve Cardiac Function in Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuejiang Liu (Other)
Responsible Party: Sponsor-Investigator, Yuejiang Liu, Associate Professor, Southeast University, China
Organization: Southeast University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: glncardio001
Record Dates: First submitted 2013-02-04; First posted 2013-02-20 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatic Heart Disease; Coronary Heart Disease
Keywords: Glutamine; Cardiosurgery; Cardiopulmonary bypass; Cardiac function; Recovery
MeSH Terms: conditions — Rheumatic Heart Disease; Coronary Disease | interventions — Glutamine; alanylglutamine; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Experimental): 20% N(2)-L-alanyl-L-glutamine 0.4g/kg(2ml/kg) mixed with compound amino acid (10ml/kg)(volume ratio=1:5).Intravenous injection twice (24 hours、1 hour before operation).
  Interventions: Drug: Glutamine
- Ringer's solution (Placebo Comparator): Ringer's solution 12ml/kg. Intravenous injection twice (24 hours、1 hour before operation).
  Interventions: Drug: Ringer's solution

INTERVENTIONS:
Drug: Glutamine — 20% N(2)-L-alanyl-L-glutamine 0.4g/kg(2ml/kg) mixed with compound amino acid (10ml/kg).Intravenous injection twice (24 hours、1 hour before operation). Injection rate = 6ml/kg/h
  Other Names: Dipeptiven (N(2)-L-Alanine L-Glutamine dipeptide)
  Arms: Glutamine
Drug: Ringer's solution — Ringer's solution 12ml/kg. Intravenous injection twice (24 hours、1 hour before operation). Injection rate = 6ml/kg/h.
  Arms: Ringer's solution

SUMMARY:
In view of the lack of large-scale clinical study and potent evidence-based medicine, the investigators designed a randomized, double-blind, placebo-controlled study to ascertain whether preoperative intravenous administration with glutamine can improve the postoperative cardiac function and prognosis of adult patients undergoing cardiac surgery. The investigators want to detect the levels of myocardial protein O-GlcNAc modification and HSP70 expression, changes in sensitive indicators of myocardial injury, systemic inflammatory reaction and oxidative stress levels, and to examine the correlation between these changes and Clinical manifestations. The ultimate goal of the study is to explore a new way for clinical myocardial protection.

DETAILED DESCRIPTION:
Cardiosurgery is mostly done under cardiopulmonary bypass. However, the cardiopulmonary bypass and the later recovery of spontaneous circulation, a cardiac ischemia / reperfusion process, may cause myocardial damage and affect cardiac function as well as prognosis.

Glutamine, an amino acid abundant in the human body, plays an important role in the regulation of metabolism and immune cells and the protection of organs. Relative lack of glutamine is reported during stress or serious illness. Animal studies have confirmed that pretreatment with glutamine has a protective effect on the heart, liver, kidney and other organs post ischemia / reperfusion injury. It is also established that glutamine exerts myocardial protection mainly by activating hexosamine biosynthetic pathway, increasing intracellular O-GlcNAc protein modification and expression of heat shock protein 70 (HSP70), starting the protective reaction in the body, improving the function of myocardial cells, and inhibiting the release of inflammatory cytokines and oxidative stress levels. Besides, clinical studies have shown that at the perioperative stage glutamine has a protective effect on cardiac function of the patients treated with pump coronary artery bypass surgery.

The purpose of this study is to ascertain whether preoperative intravenous administration with glutamine (as compared with control group) can improve the postoperative cardiac function and prognosis of adult patients undergoing cardiac surgery and reduce inflammatory response and oxidative stress levels of the body. The correlation between Clinical manifestations and expression of myocardium O-GlcNAc and HSP70 will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with coronary artery disease or rheumatic heart disease accepted cardiosurgery under cardiopulmonary bypass

Exclusion Criteria:

* ejection fraction(EF)<50%
* Preoperative support with intra-aortic balloon pump(IABP)
* Hepatosis
* Renal dysfunction
* Myocardial infarction attack within 3 months
* Emergency operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
perioperative changes of Cardiac Index (CI) | postanescesia before surgery, 2, 20 hours after cardiopulmonary bypass (CPB)
  For each patient,a Swan-Ganz catheter will be inserted after anesthesia induction.CI and other values of hemodynamics will be measured.

SECONDARY OUTCOMES:
Troponin I(cTnI) | postanescesia before surgery, 6, 20 hours after CPB
  CTnI is a sensitive indicator of myocardial damage.
Brain Natriuretic Peptide (BNP) | postanescesia before surgery, 6, 20 hours after CPB
  BNP is a sensitive indicator of cardiac dysfunction.
Systemic inflammation | postanescesia before surgery, 2, 20 hours after CPB
  Blood levels of Interleukin-6（IL-6）、Tumor Necrosis Factor（TNF-a） and Malondialdehyde (MDA) will be measured.
Heart issue HSP-70 | 20 minutes after CPB
  A mass of heart tissue (a part of right auricle of heart,weigh about 50mg) will be cut 20 minutes after CPB for the measurements.
Heart issue O-GlcNAc | 20 minutes after CPB
  The same mass of heart tissue described above will be used for the measurements.
Recovery index | Date of surgery until date of hospital discharge (an expected average of 2 weeks)
  Recovery index include duration of mechanical ventilation、duration of ICU stay、duration of hospital stay、adverse event and mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China